CLINICAL TRIAL: NCT07239141
Title: Estimation of the Non-Inferiority of the Laringocel® Videolaryngoscope Compared With the C-MAC D-BLADE (Karl Storz®) for First-Attempt Intubation in Adult Patients Undergoing Elective Surgery
Brief Title: Two Video Laryngoscopes (Laringocel® and C-MAC®) for First-Attempt Intubation in Adults Undergoing Elective Surgery
Acronym: LARINGOCOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Zamudio (Other)
Responsible Party: Sponsor-Investigator, Mario Zamudio, University professor with a master's degree in clinical epidemiology, Universidad de Antioquia
Organization: Universidad de Antioquia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IN29-2025
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Airway Management; Intubation, Endotracheal
Keywords: Videolaryngoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: the person who generated the randomization sequence is independent from patient recruitment, intervention, and outcome assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laringocel (Experimental): Participants in this group will undergo orotracheal intubation using the Laringocel videolaryngoscope
  Interventions: Device: Laringocel® videolaryngoscope
- C-MAC D-Blade (Active Comparator): Participants in this group will undergo orotracheal intubation using the C-MAC D-Blade video laryngoscope (Karl Storz).
  Interventions: Device: C-MAC® D-Blade videolaryngoscope

INTERVENTIONS:
Device: Laringocel® videolaryngoscope — Orotracheal intubation performed with a hyperangulated Laringocel® videolaryngoscope by board-certified anesthesiologists who have completed a validated learning curve (CUSUM).
  Participants will undergo general anesthesia with adequate neuromuscular relaxation. The type and dose of anesthetic drugs will be determined by the attending anesthesiologist, ensuring at least an effective dose equivalent to ED95. If succinylcholine is used, intubation will be performed 45 seconds after administration; for cisatracurium, after 4 minutes; and for vecuronium or rocuronium, after 2 minutes.
  Arms: Laringocel
Device: C-MAC® D-Blade videolaryngoscope — Orotracheal intubation performed with a hyperangulated C-MAC® D-Blade videolaryngoscope (Karl Storz®) by board-certified anesthesiologists who have completed a validated learning curve (CUSUM).
  Participants will undergo general anesthesia with adequate neuromuscular relaxation. The type and dose of anesthetic drugs will be determined by the attending anesthesiologist, ensuring at least an effective dose equivalent to ED95. If succinylcholine is used, intubation will be performed 45 seconds after administration; for cisatracurium, after 4 minutes; and for vecuronium or rocuronium, after 2 minutes.
  Arms: C-MAC D-Blade

SUMMARY:
This study will test two video laryngoscopes that help doctors place a breathing tube during surgery. A breathing tube is needed for people who receive general anesthesia so they can breathe safely. Video laryngoscopes use a small camera to give a better view of the throat and vocal cords, which may help the tube go in on the first try.

The purpose of this research is to find out if a Colombian device called Laringocel® works as well as the widely used international device C-MAC D-Blade® (Karl Storz). If Laringocel® performs similarly, it could be a more affordable option for hospitals with limited resources.

252 adults (126 in each group) who need elective surgery at Alma Máter Hospital de Antioquia (Medellín, Colombia) will take part. Each participant will be randomly assigned, like flipping a coin, to have their breathing tube placed with either Laringocel® or C-MAC D-Blade®. Only trained anesthesiologists will perform the procedure.

The study will look at:

Main goal: how often the tube goes in correctly on the first attempt.

Other goals: overall success within 3 attempts, how well the airway is seen, how long the intubation takes, how satisfied the doctor is with the device, and possible side effects such as sore throat, dental injury, or oral injury.

Participation will not change the usual care people receive during anesthesia. Both devices are already approved for clinical use. Risks are the same as with any standard intubation, and participants will be checked after surgery for any problems.

By comparing these two devices, researchers hope to learn if Laringocel® can provide safe and effective intubation at lower cost, improving access to advanced airway tools.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients scheduled for elective surgery under general anesthesia
* Patients requiring single-lumen orotracheal intubation
* Patients compliant with the anesthetic indication and standard preoperative fasting requirements

Exclusion Criteria:

* Patients with an anticipated difficult airway (more than two anatomical risk factors for difficult airway)
* Patient refusal to participate in the study via informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
First-attempt orotracheal intubation success | During the intubation procedure (intraoperative, immediately after induction of anesthesia)
  Proportion of participants with successful tracheal intubation on the first attempt, defined as correct placement of the endotracheal tube confirmed by continuous capnography. A successful attempt is one in which the videolaryngoscope is introduced and removed only once, without requiring a second attempt, device change, or external assistance.

SECONDARY OUTCOMES:
Overall orotracheal intubation success within three attempts | During the intubation procedure (intraoperative, immediately after induction of anesthesia)
  Proportion of participants with successful tracheal intubation within a maximum of three attempts using the assigned videolaryngoscope, defined as correct tube placement confirmed by continuous capnography.
Percentage of Glottic Opening (POGO) score | During the intubation procedure (intraoperative, immediately after induction of anesthesia)
  Continuous measure from 0 to 100% estimating the visible portion of the vocal cords during videolaryngoscopy. Higher values indicate a better glottic view. Mean POGO scores will be compared between intervention groups.
Fremantle score | During the intubation procedure (intraoperative, immediately after induction of anesthesia).
  Ordinal scale combining the best laryngeal view obtained (Full, Partial, None) and ease of intubation (1 = easy, 2 = modified, 3 = impossible). Lower scores indicate easier intubation.
Intubation time | During the intubation procedure (intraoperative, immediately after induction of anesthesia)
  Time in seconds from insertion of the videolaryngoscope into the mouth until confirmation of successful tracheal tube placement by capnography.
Operator satisfaction | Immediately after the intubation procedure (intraoperative period)
  Mean score of four items on a 5-point Likert scale evaluating technical ease, physical comfort, overall satisfaction, and willingness to reuse the device (1 = very satisfied, 5 = not satisfied).
Team situation awareness (SAGAT method) | Immediately after the intubation procedure (intraoperative period)
  Assessed by an external observer using the Situation Awareness Global Assessment Technique (SAGAT). Binary responses to three questions representing perception, comprehension, and projection of the situation.
Adverse events related to intubation | One hour after extubation (post-anesthesia care unit or intensive care unit)
  Proportion of participants presenting sore throat, dental injury, or visible mucosal/oropharyngeal lesions after extubation, assessed by direct examination and participant report.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Alma Máter de Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the published results will be shared. This will include demographic data, airway characteristics, and outcome variables used in the analyses. A data dictionary will accompany the dataset.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The de-identified individual participant data and supporting documentation will be available after the study is completed and the main results are published. Data will remain accessible for 5 years. After this period, requests will be evaluated on a case-by-case basis, depending on data storage conditions and the status of ethical approval.
Access Criteria: Access will be granted to qualified researchers with methodologically sound proposals for secondary analyses that align with the study objectives or advance research in airway management. Proposals will be reviewed by the Principal Investigator and the Institutional Ethics Committee of Hospital Alma Máter de Antioquia. Approved applicants must sign a data access agreement outlining confidentiality, data security, and publication terms. Requests should be sent to gabriel.munoz@udea.edu.co.

REFERENCES:
- [Background] Sotres-Ramos D, Almendra-Arao F, Anguiano-Mondragon E. A New Method for the Comparison of Powers of Noninferiority Exact Tests for the Difference of Proportions. Ther Innov Regul Sci. 2014 Sep;48(5):592-600. doi: 10.1177/2168479014523005. PMID 30231446
- [Background] Mort TC. Emergency tracheal intubation: complications associated with repeated laryngoscopic attempts. Anesth Analg. 2004 Aug;99(2):607-13, table of contents. doi: 10.1213/01.ANE.0000122825.04923.15. PMID 15271750
- [Background] Zhang J, Jiang W, Urdaneta F. Economic analysis of the use of video laryngoscopy versus direct laryngoscopy in the surgical setting. J Comp Eff Res. 2021 Jul;10(10):831-844. doi: 10.2217/cer-2021-0068. Epub 2021 Apr 27. PMID 33904779
- [Background] Heidegger T. Management of the Difficult Airway. N Engl J Med. 2021 May 13;384(19):1836-1847. doi: 10.1056/NEJMra1916801. No abstract available. PMID 33979490
- [Background] Piaggio G, Elbourne DR, Pocock SJ, Evans SJ, Altman DG; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: extension of the CONSORT 2010 statement. JAMA. 2012 Dec 26;308(24):2594-604. doi: 10.1001/jama.2012.87802. PMID 23268518
- [Background] Aziz MF, Abrons RO, Cattano D, Bayman EO, Swanson DE, Hagberg CA, Todd MM, Brambrink AM. First-Attempt Intubation Success of Video Laryngoscopy in Patients with Anticipated Difficult Direct Laryngoscopy: A Multicenter Randomized Controlled Trial Comparing the C-MAC D-Blade Versus the GlideScope in a Mixed Provider and Diverse Patient Population. Anesth Analg. 2016 Mar;122(3):740-750. doi: 10.1213/ANE.0000000000001084. PMID 26579847
- [Background] Hansel J, Rogers AM, Lewis SR, Cook TM, Smith AF. Videolaryngoscopy versus direct laryngoscopy for adults undergoing tracheal intubation. Cochrane Database Syst Rev. 2022 Apr 4;4(4):CD011136. doi: 10.1002/14651858.CD011136.pub3. PMID 35373840
- [Background] Apfelbaum JL, Hagberg CA, Connis RT, Abdelmalak BB, Agarkar M, Dutton RP, Fiadjoe JE, Greif R, Klock PA, Mercier D, Myatra SN, O'Sullivan EP, Rosenblatt WH, Sorbello M, Tung A. 2022 American Society of Anesthesiologists Practice Guidelines for Management of the Difficult Airway. Anesthesiology. 2022 Jan 1;136(1):31-81. doi: 10.1097/ALN.0000000000004002. PMID 34762729
- [Background] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488

DOCUMENTS (3):
  • Study Protocol (2025-09-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT07239141/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT07239141/SAP_001.pdf
  • Informed Consent Form (2025-09-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT07239141/ICF_002.pdf